CLINICAL TRIAL: NCT01426724
Title: Effects of Active Form of Vitamin D on Renal Blood Flow, Glomerular Filtration Rate, Proteinuria and Inflammation in Patients With Chronic Kidney Disease and Hyperparathyroidism
Brief Title: Effects of Vitamin D on Renal Blood Flow, Proteinuria and Inflammation in Patients With Chronic Kidney Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficult to enroll eligible subjects.
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Kambiz Kalantarinia, MD, Principal Investigator, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 15043
Record Dates: First submitted 2011-08-29; First posted 2011-08-31 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Chronic Kidney Disease; Secondary Hyperparathyroidism
Keywords: Vitamin D; Chronic Kidney Disease; Hyperparathyroidism; Renal Blood Flow; Proteinuria; Inflammation; Renin Angiotensin System
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperparathyroidism, Secondary; Hyperparathyroidism; Proteinuria; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Contrast Enhanced Ultrasonography — Definity microbubbles will be infused intravenously at a rate of 2mL/min. contrast enhanced images of the kidneys will be obtained during the infusion and following the destruction of microbubbles within the kidney tissue with ultrasound to measure renal blood flow two times within a 90 day (plus or minus 10 day) window

SUMMARY:
Active forms of vitamin D and its analogs are used to treat elevated parathyroid hormone levels and bone disease in chronic kidney disease (CKD). More recent animal and human studies suggest that treatment with vitamin D may be associated with reduction of inflammation and urinary protein loss as well as reduction the activity of the renin angiotensin system (RAS) in addition to its effects on the bone metabolism. The investigators of this study have used the new technique of contrast enhanced ultrasound (CEU) to measure the flow of blood to the kidney in other human studies. In this study, the investigators will investigate if 3 month of treatment with an active form of vitamin D in individuals with kidney disease and high parathyroid hormone levels would reduce protein loss in the urine. The investigators will also look at the potential changes in blood flow to the kidney using CEU, kidney function (GFR), inflammation and activity of RAS in response to treatment with active form of vitamin D. Finally, they will examine the association between reduction of protein loss in the urine as shown in other studies with any of the other factors measured (e.g, change in blood flow or inflammation).

DETAILED DESCRIPTION:
Screening visit, (Day 1) Most subjects will be contacted during their visit to the Kidney Center Clinic. In some cases, subjects are identified a few days after their visit with their nephrologists and once their laboratory results are available. If a subject is eligible for participation in the study, screening visit will occur at the Nephrology Clinical Research Center located right next to the Kidney Center Clinic. The following will occur during the screening visit,

1. Inclusion and exclusion criteria will be reviewed
2. Details of the study procedures will be reviewed with the subject
3. Informed consent is signed and the subjects will be enrolled in the study.
4. A physical exam will be performed.
5. Vital Signs will be taken (blood pressure and heart rate)
6. A urine pregnancy test will be performed for women of child bearing age. If positive subjects will be excluded.
7. If a urine test for proteinuria is not ordered at the clinic visit by subjects' nephrologist, a urine sample will be collected and sent to the laboratory for urine creatinine and urine protein.
8. Subjects will be asked to present to the CRU within one week of their screening visit in the morning.
9. Subjects will be asked not to start vitamin D pills prescribed by their nephrologists until after completing study visit 2 procedures.

Visit 2 (Day 2 - 7).

1. Eligibility will be reviewed.
2. A physical exam will be performed.
3. Vital Signs will be taken (blood pressure and heart rate)
4. A urine sample will be collected and will be tested for,

   * Urine creatinine (baseline)
   * Urine protein (baseline)
   * Urine hcg to check for pregnancy in women of child bearing age
   * Urinalysis
5. Subjects with a positive urine pregnancy test will be excluded
6. A large bore intravenous catheter will be placed in a peripheral vein for the purpose of infusion of Definity and will be locked with heparin.
7. Blood samples will be collected at the time of IV catheter placement. These samples will be checked for baseline concentrations of ,

   * IL-1, IL-6, CRP, and TNF-alpha
   * Plasma renin activity and serum aldosterone
   * Basic metabolic panel
   * Serum albumin
8. Subjects will be placed on a continuous cardiac monitor and pulse oximetry. If oxygen saturation is <90% the subject will be excluded
9. Subjects will need to lie in bed on their back and remain in bed until the test procedures are completed (may be up to use a bedside commode).
10. Resting ultrasonography will be performed on both kidneys to determine kidney volume, and Doppler studies will be done.
11. Color Doppler from the subcostal view will be performed to rule out the possibility of intracardiac shunts. These individuals will be excluded from the study.
12. The Definity vial will be placed at room temperature before being used. It will be activated after shaking the vial using Vialmax for 45 seconds. It will be used immediately after activation.
13. 1.3 ml of Definity will be mixed in 30 ml of preservative free saline. Infusion of Definity into a peripheral vein will be started at 2 ml/min and titrated for optimal image quality (not to exceed 10 ml/min at any time).
14. To assess optimal microbubble concentration based upon video intensity, ultrasound images of the left ventricle will be obtained and used as the control. Microbubble administration will then be titrated accordingly but not to exceed 10 ml/min at any time.
15. Baseline contrast ultrasound imaging of right kidney will be performed using Power Modulation imaging with low mechanical index (MI) of 0.1.
16. One to four impulses with high MI of 1.0 will be used to destruct the microbubbles and then imaging of the kidney with low MI (0.1) will continue for several seconds to a few minutes. Infusion of Definity will stop at this point.
17. During the administration of Definity, vital signs including heart rate and pulse oximetry will be obtained continuously
18. Study subjects will stay in CRU for 30 minutes of observation (continuous ECG monitoring and frequent blood pressure, pulse, respiratory rate and oxygen saturation monitoring will continue during this period.
19. A urine sample will be collected for urinalysis.
20. Subjects will be discharged home.
21. At the time of discharge each subject will be asked to start taking the active vitamin D pill prescribed by their nephrologists. They will be asked to inform us if they stop their medication for any reason within the next three months.
22. Subjects will be asked to not to start any new blood pressure medications during the time of the study. They will be asked to contact us if a change is made to any of their medications.
23. Between 48 - 72 hours after discharge from CRU subjects will be contacted to assess for adverse events.
24. After three months of treatment with one form of vitamin D, the subjects will return to the CRU for the following procedures,

    Visit 3 (day 83 - 107) 90 ± 10 days after visit 1
25. Eligibility will be reviewed.
26. A physical exam will be performed.
27. Vital Signs will be taken (blood pressure and heart rate)
28. A urine sample will be collected and will be tested for,

    * Urine hcg to check for pregnancy in women of child bearing age
    * Urine creatinine (end of study)
    * Urine protein (end of study)
    * Urinalysis
29. Women with a positive pregnancy test will be excluded
30. A large bore intravenous catheter will be placed in a peripheral vein for the purpose of infusion of Definity and will be locked with heparin.
31. Blood samples will be collected at the time of IV catheter placement. These samples will be checked for baseline concentrations of ,

    * IL-1, IL-6, CRP, and TNF-alpha
    * Plasma renin activity and serum aldosterone
    * Basic metabolic panel
    * Serum albumin
    * Serum calcium, phosphorus and intact PTH concentrations, unless done as standard of care within a week of end of study visit.
32. Steps 6 - 20 mentioned above will be repeated.
33. Between 48 - 72 hours after discharge from the CRU subjects will be contacted by phone to assess for potential adverse events.
34. Study procedures will end at this time.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (ages 18 - 75 years)
2. A diagnosis of chronic kidney disease (CKD) with a glomerular filtration rate (GFR) in the range of 20 - 60 ml/min/1.73 m2.
3. Proteinuria confirmed at least twice by one of the following (at least one sample within the last 6 months),

   * 24-hour urine protein excretion of at least 150 mg/day OR
   * spot urine protein to creatinine ratio (PCR) of greater than 0.15 OR
   * spot urine albumin to creatinine ratio (ACR) greater than 100 mg/g
4. A recent diagnosis of secondary hyperparathyroidism of renal origin by the patient's nephrologist scheduled for treatment with an active from of vitamin D.
5. Available results for serum intact parathyroid hormone (iPTH), calcium and phosphorus within 6 months from the study enrollment date.
6. Treatment with a stable dose of an angiotensin receptor blocker (ARB), angiotensin converting enzyme inhibitor (ACE-I) or rennin inhibitor within the last 2 months before enrollment in the study.

Exclusion Criteria:

1. GFR less than 20 or greater than 60 ml/min/1.73 m2.
2. Treatment with an active form of vitamin D, including Calcitriol (Rocaltrol), Paricalcitol (Zemplar) and Doxercalciferol (Hectorol) within the last 3 months.
3. Need for renal replacement therapy within the next three months.
4. History of any organ transplantation requiring immunosuppressive therapy.
5. Chronic treatment with anti-inflammatory agents including NSAIDs, steroids or cytotoxic agents.
6. Diagnoses of primary or tertiary hyperparathyroidism.
7. Serum intact parathyroid hormone (PTH) concentration greater than 250 pg/mL.
8. Serum calcium greater than 10.4 mg/dL.Serum phosphorous greater than 5 mg/dL.
9. Active malignancy.
10. History of systemic inflammatory diseases such as, systemic lupus, rheumatoid arthritis or vasculitis.
11. History of pulmonary hypertension, intracardiac shunt or unstable cardiopulmonary disease.
12. Women who are pregnant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in proteinuria compared to baseline as determined by spot urine protein to creatinine ratio (PCR) | Subjects must be on Vitamin D for 90 days (plus or minus 10 days)
  The pre to post-intervention change in urinary protein to creatinine ratio (PCR) will be analyzed either by way of the common paired Students t-test or the by way of paired Wilcoxon test. The paired Student t-test will be utilized if the measurements of the pre to post-intervention change in PCR are normally distribution, otherwise the ranked based paired Wilcoxon test will be utilized.

SECONDARY OUTCOMES:
Change in renal blood flow compared to baseline as determined by contrast enhanced ultrasound. | Subjects must be on Vitamin D for 90 days (plus or minus 10 days)
  Baseline RBF will be measured using contrast enhanced ultrasound. subjects will be treated with one of the active forms of vitamin D for 90 days. Measurement of RBF usinf CEU will be repeated. Same statisticak methods will be used for this outcome as the primary outcome of the study.
Association between changes from baseline in PCR and RBF | Subjects must be on Vitamin D for 90 days (plus or minus 10 days)
  We will examine whether the pre-intervention to post-intervention changes in PCR were associated with changes in either renal blood flow. Spearman rank correlations and Spearman partial-rank correlations will be utilized to examine possible associations. With regard to hypothesis testing, the null hypothesis of no association will be rejected based on a p≤0.05 decision rule.
Association between changes from baseline in PCR and GFR | Subjects must be on Vitamin D for 90 days (plus or minus 10 days)
  We will examine whether the pre-intervention to post-intervention changes in PCR were associated with changes in GFR. Spearman rank correlations and Spearman partial-rank correlations will be utilized to examine possible associations. With regard to hypothesis testing, the null hypothesis of no association will be rejected based on a p≤0.05 decision rule.
Association between changes from baseline in PCR and concentration of biomarkers of inflammation | Subjects must be on Vitamin D for 90 days (plus or minus 10 days)
  We will examine whether the pre-intervention to post-intervention changes in PCR were associated with changes in CRP, IL-1, IL-6, or TNF-alpha. Spearman rank correlations and Spearman partial-rank correlations will be utilized to examine possible associations. With regard to hypothesis testing, the null hypothesis of no association will be rejected based on a p≤0.05 decision rule.
Association between changes from baseline in PCR and activity of the renin angiotensin system. | Subjects must be on Vitamin D for 90 days (plus or minus 10 days)
  We will examine whether the pre-intervention to post-intervention changes in PCR were associated with changes in plasma renin-activity and plasma aldosterone concentration. Spearman rank correlations and Spearman partial-rank correlations will be utilized to examine possible associations. With regard to hypothesis testing, the null hypothesis of no association will be rejected based on a p≤0.05 decision rule.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States